CLINICAL TRIAL: NCT07242547
Title: A Phase II Clinical Trial of Tarlatamab as Maintenance Treatment After Sequential Chemo-radiotherapy for Limited Stage SCLC Patients Not Eligible for Concurrent Chemo-radiotherapy
Brief Title: Study of Tarlatamab as Maintenance Treatment After Chemo-radiotherapy for Limited Stage SCLC Patients
Acronym: MERLIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 24/01_MERLIN; 2024-515201-26-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Limited-stage Small-cell Lung Cancer; Carcinoma, Small Cell Lung; Respiratory Tract Neoplasms; Thoracic Neoplasms
Keywords: Non small cell lung cancer; Tarlatamab; Maintenance treatment; Antineoplastic Agents; Chemo-radiotherapy; Immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma; Respiratory Tract Neoplasms; Thoracic Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Maintenance treatment (Experimental): Patients will be enrolled in the trial after receiving sequential chemo-radiotherapy, if there is no progression disease, patients will receive tarlatamab maintenance treatment.
  Patients will receive maintenance with Tarlatamab IV until disease progression unacceptable toxicity, patient or physician decision to discontinue or death.
  Interventions: Drug: Tarlatamab

INTERVENTIONS:
Drug: Tarlatamab — Patients will be enrolled in the trial after receiving sequential chemo-radiotherapy, if there is no progression disease, patients will receive tarlatamab maintenance treatment.
  Patients will receive maintenance with tarlatamab IV until disease progression unacceptable toxicity, patient or physician decision to discontinue or death.
  Patients who still benefit from the drug treatment at the end of the study or at early termination of the clinical trial, will continue receiving the drug until progression disease.
  Other Names: Imdelltra

SUMMARY:
This is an open-label, phase II, exploratory and multi-centre clinical trial. 37 Limited stage SCLC patients not eligible for concurrent chemo-radiotherapy will be enroll.

Patients will be enrolled in the trial after receiving sequential chemo-radiotherapy, if there is no progression disease, patients will be treated with maintenance Tarlatamab.

Patients will receive maintenance with Tarlatamab IV until disease progression unacceptable toxicity, patient or physician decision to discontinue or death.

The primary objective is to evaluate the Progression free survival (PFS).

Patient accrual is expected to be completed within 2 years. Treatment and follow-up are expected to extend the study duration to a total of 5 years. Patients will be followed for 2 years after enrollment. The study will end once survival follow-up has concluded.

DETAILED DESCRIPTION:
The study MERLIN is a phase II clinical trial intending to enroll 37 patients, who will receive will receive Tarlatamab as maintenance treatment.

This is an open-label, phase II, exploratory and multi-centre clinical trial. Limited stage SCLC patients not eligible for concurrent chemo-radiotherapy will be selected.

Patients will be enrolled in the trial after receiving sequential chemo-radiotherapy, if there is no progression disease, patients will be treated with maintenance Tarlatamab.

Patients will receive maintenance with Tarlatamab IV until disease progression unacceptable toxicity, patient or physician decision to discontinue or death.

For all patients, tumor response data collection will continue until disease progression, even if the patient stops study treatment prior to disease progression.

Patients who still benefit from the drug treatment at the end of the study or at early termination of the clinical trial, will continue receiving the drug until progression disease.

The primary objective is to evaluate the Progression free survival (PFS) in the intent-to-treat population. Progression free survival (PFS) defined as the time from enrollment to the date of the first documentation of disease progression according to RECIST 1.1 or death from any cause, whichever is earlier

Patient accrual is expected to be completed within 2 years. Treatment and follow-up are expected to extend the study duration to a total of 5 years. Patients will be followed for 2 years after enrollment. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented new diagnosis of LS-SCLC by histology or cytology from brushing, washing, or needle aspiration. Mixed tumors are not eligible.
* Patients who:

  1. were treated with sequential chemo-radiotherapy
  2. were treated only with chemotherapy
* Have at least one lesion that meets criteria for being measurable or non-measurable, as defined by RECIST 1.1.
* Has completed chemo-radiation or chemotherapy alone without progression of disease per RECIST v1.1
* Be male or female ≥18 years of age inclusive, on the day of signing informed consent.
* Have a life expectancy of at least 3 months from the study start.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 within 7 days prior to the first dose of study intervention.
* Toxicities attributed to chemo-radiotherapy treatment have to be resolved to grade ≤1, unless otherwise specified.
* No clinically significant electrocardiogram (ECG) findings
* Correct pulmonary function without oxygen supplementation
* Have voluntarily agreed to participate by giving written consent for the study prior to any specific protocol procedures.
* Have adequate organ function (hematological and biochemistry parameters).

Exclusion Criteria:

* Patients expected to require any other form of radiation therapy for LS-SCLC as concurrent radiotherapy.
* Extensive-stage SCLC (ES-SCLC) or any previous diagnosis of transformed non-small cell lung cancer. Mixed tumors (SCLC-NSCLC) are not eligible.
* Has known history of, or active, neurologic paraneoplastic syndrome of autoimmune nature.
* Has had major surgery within 4 weeks prior to first dose of study interventions.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has known history of a second malignancy other than SCLC, unless potentially curative treatment has been completed with no evidence of malignancy for at least 3 years since the initiation of that therapy.
* Uncontrolled intercurrent active infection at the time of enrollment requiring systemic therapy.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* History of solid organ transplantation.
* Myocardial infarction and/or symptomatic congestive heart failure (New York Heart Association >class II) within 6 months prior to first dose of study treatment.
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has a known history of Hepatitis B or known active Hepatitis C virus infection.
* Has a known history of active tuberculosis.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has serious nonhealing wound, ulcer, or bone fracture within 28 days before first dose of study intervention.
* Female subjects of childbearing potential unwilling to use protocol specified method of contraception during treatment and for an additional 60 days after the last dose of study treatment.
* Female subjects who are breastfeeding or who plan to breastfeed while on study through 60 days after the last dose of study treatment.
* Female subjects planning to become pregnant or donate eggs while on study through 60 days after the last dose of study treatment.
* Female subjects of childbearing potential with a positive pregnancy test assessed at screening by a highly sensitive serum pregnancy test.
* Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence or use contraception during treatment and for an additional 60 days after the last dose of study treatment.
* Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom during treatment and for an additional 60 days after the last dose of study treatment.
* Subject has known sensitivity to any of the products or components to be administered during dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of enrollment until the date of last follow up, assessed up to 24 months.
  Efficacy of Tarlatamab as maintenance treatment assessed by progression free survival Progression-free survival, defined as the time from enrollment to the date of the first documentation of disease progression according to Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) or death from any cause, whichever is earlier. Progression is defined using RECIST v1.1, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
Objective response rate (ORR) | From the date of enrollment to the date of last follow up, assessed up to 24 months
  ORR: Describe the efficacy of Tarlatamab as maintenance treatment as assessed by objective response rate (ORR) Investigator-assessed ORR, defined as a confirmed complete response (CR) plus partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1). According to RECIST 1.1, a complete response is the disappearance of all target lesions, and a partial response is defined as at least a 30% decrease in the sum of the target lesions.
Overall Survival (OS) | From the date of enrollment to 6 months, 1 and 2 years
  OS at 6 months and 1 and 2 years, defined as the time from enrollment to the date of death from any cause
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | From the subject's written consent to participate in the study through 90 days after the final administration of the drug.
  Occurrence and severity of adverse events, with severity determined by NCI CTCAE v5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — President of Grupo Español de Cáncer de Pulmón
Locations (20):
- Spain (20):
  - Hospital General Universitario de Albacete, Albacete, Albacete
  - Hospital General Universitario Dr. Balmis de Alicante, Alicante, Alicante
  - Hospital General Universitario de Elche, Elche, Alicante
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Fundació Althaia, Manresa, Barcelona
  - Hospital de Basurto, Bilbao, Bizkaia
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid, Madrid
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital Regional de Málaga, Málaga, Málaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Hospital Santa Maria Mai - Complexo Hospitalario Universitario Ourense, Ourense, Ourense
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital General Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org